CLINICAL TRIAL: NCT01333319
Title: The Role of Biomarkers in the Early Detection of Acute Kidney Injury Induced by Liver Transplantation : an Observational Analysis.
Brief Title: The Role of Biomarkers in the Early Detection of Acute Kidney Injury Induced by Liver Transplantation
Acronym: KILT
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: KILT1
Record Dates: First submitted 2011-04-08; First posted 2011-04-11 (Estimated); Last update posted 2023-01-27 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Injury
Keywords: liver transplantation; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Renal dysfunction is a major risk factor for poorer outcome after liver transplantation. Nevertheless, mechanisms of renal dysfunction in liver transplant recipients are not clearly understood. Calcineurin inhibitors are generally perceived as the most important cause; however the liver transplant procedure itself represents a major surgical / hemodynamic / inflammatory trauma that - on its own - can cause renal dysfunction. Creatinine and creatinine clearance are late markers of acute kidney injury and changes in these parameters occur only after substantial injury has already occurred. Even a stable creatinine does not exclude structural kidney damage.

A series of new markers of tissue injury have been identified and have the potential to identify acute kidney injury better and earlier than creatinine and creatinine clearance. The aim of this study is to determine whether and how liver transplantation affects these urinary and plasma biomarkers and to study whether the changes in these biomarkers may predict later changes in standard functional parameters (creatinine and creatinine clearance). For this purpose, the urinary and plasma biomarkers, together with creatinine, will be determined serially during the different phases of the liver transplant process and daily until day 5 after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years

Exclusion Criteria:

* Younger than 18 years old
* Combined organ transplants
* Dialysis dependent prior to liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the University Hospitals Leuven listed on the Eurotransplant waiting list for liver transplantation and undergoing a liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-12; Primary Completion 2015-06 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Biomarkers in urine and plasma | First 5 days post transplantation

SECONDARY OUTCOMES:
Creatinine change | First 5 days post transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Pirenne, MD, PhD, Principal Investigator — Abdominal Transplant Surgery, University Hospitals Leuven, KULeuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium